CLINICAL TRIAL: NCT04538456
Title: Understanding the Physical, Social and Psychological Impact of COVID-19 on Frail and Shielded Lung Cancer Patients
Brief Title: Impact of COVID-19 on Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp189
Record Dates: First submitted 2020-09-01; First posted 2020-09-04 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer; PROM; Covid19; Psychological
MeSH Terms: conditions — Lung Neoplasms; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- used electronic Patient Reported Outcome Measures: Lung cancer patients who have used the electronic Patient Reported Outcome Measures system before and after COVID-19 lock down or new patients who have completed their first electronic Patient Reported Outcome Measures after COVID-19 lock down.
  Interventions: Other: questionnaire and optional interview
- never used electronic Patient Reported Outcome Measures: Lung cancer patients who have never completed electronic Patient Reported Outcome Measures.
  Interventions: Other: questionnaire and optional interview

INTERVENTIONS:
Other: questionnaire and optional interview — Participants will be sent an online or paper questionnaire. If participants have expressed an interest in taking part in an interview, they may be contacted by a member of the research team. The interviews will be conducted over the phone at time suitable for the participant. There will be no study specific hospital visits.

SUMMARY:
During the COVID-19 pandemic, people's lives have changed dramatically. People with lung cancer who are shielding may have been particularly affected as they may be unable to carry out many of their normal daily activities, such as grocery shopping and exercise, and are unable to interact with friends and family. People with lung cancer will also have experienced some changes to the clinical services available to them at The Christie. Using a questionnaire and interviews, the investigators want to understand patient experiences of the changes in their daily lives and the changes to their clinical care. This will help us to see if people with lung cancer need any additional support services or if there are any changes the investigators can make to clinical services to improve patient experiences. Eligible patients will be any lung cancer patients receiving current treatment or in active follow up.

DETAILED DESCRIPTION:
The COVID-19 pandemic, declared by the World Health Organisation (WHO) on 11 March 2020, has managed to dramatically change all of our lives in just a few short months. Due to the unprecedented demand to protect the National Health service (NHS), on 23 March 2020 the United Kingdom (UK) government initiated a lock down, imposing wide-ranging restrictions on freedom of movement. Cancer services have been being particularly impacted across the country.

Around 48,000 patients are newly diagnosed with lung cancer in the UK each year. Those who require active treatment may be offered radiotherapy, systemic anticancer therapy including chemotherapy, targeted therapy or immunotherapy, or a combination of both. A recent document published by Public Health England(PHE) has classified lung cancer patients receiving any of these treatments as 'extremely vulnerable.' Common co-existing comorbidities such as Chronic Obstructive Pulmonary Disease (COPD) also place patients into this category. Their vulnerability may be further amplified when considering that 44% of all new lung cancer diagnoses are in people aged >75 years and a significant proportion is particularly frail. The advice from PHE for these 'extremely vulnerable' patients was to shield, meaning they should not leave their homes or attend any social gatherings, even with family or friends. Shielding unfortunately is not without its own challenges. It may prevent many patients from carrying out their daily life activities independently, limit their ability to exercise and impact their mental further. This is particularly relevant for those patients more vulnerable or frail. It would therefore be expected that these patients are likely to develop some degree of psychological distress. The act of shielding itself may be implicated in this owing to increased social isolation, upset to normal routines and general anxiety regarding COVID-19 related or other issues. In addition any change to routine lung cancer management in these patients may exacerbate this distress further. Those with underlying mental health issues are at particular risk.

During the COVID-19 pandemic both the lung cancer diagnosis and its subsequent management have been affected. These rapid changes reflected the shifting risk-benefit ratio for patients and diminished resources. Beyond modifications in treatment pathways, telephone consultations have replaced many face to face appointments in an attempt to reduce visits to hospital. The use of electronic Health tools and telemedicine has therefore suddenly come to the fore front of clinical practice.

At the Christie NHS Foundation Trust, all lung cancer patients have been given the opportunity to regularly complete electronic patient reported outcome measures routinely as part of their clinical care since December 2018. Patients are sent a text message either on the day of a new patient appointment or three days before a follow-up appointment. They are asked to complete the electronic Patient Reported Outcome Measures specifically selected for each patient's diagnosis and treatment pathway including a list of symptoms based on the Common Terminology Criteria for Adverse Events. The EuroQual-5D quality of life questionnaire is also included. This allows clinicians to review patients' symptoms before the consultation, allowing him/her to focus on the concerning symptoms and quality of life issues. Moreover, all new lung cancer patients are also screened for frailty within the Frailty Project through the electronic use of Rockwood Clinical Frailty Scale which is performed by clinicians.

ELIGIBILITY:
Inclusion Criteria:

* non-small cell lung cancer (NSCLC) or small cell lung cancer (SCLC)
* patients in active treatment or in clinical follow-up

Exclusion Criteria:

* Lung cancer patients who do not speak or understand English will not be eligible to take part in the study
* Patients under the age of 18 will be eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Additionally, participants will need to meet the criteria to be selected for one of the two cohorts of patients:
  1. Lung cancer patients voluntarily using the ePROMs platform with at least 1 assessment completed in the 6 months prior to 23 March 2020 (COVID-19 lockdown date) and 1 assessment after this date or new patients who have completed their first electronic Patient Reported Outcome Measures after 23 March 2020
  2. Lung cancer patients who have never complete electronic Patient Reported Outcome Measures data.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-04-16 (Actual); Study Completion 2022-04-16 (Actual)

PRIMARY OUTCOMES:
Physical and Social impact | baseline
  Physical and social impact will be captured by the EuroQual-5D quality of life and questions regarding patient's diagnosis and treatment pathway including a list of symptoms based on the Common Terminology Criteria for Adverse Events.
Psychological impact | baseline
  Emotional impact will be assessed using the Hospital Anxiety Depression Scale. Scores range from 0-21 for each of the two subscales (anxiety and depression), with higher scores indicating greater anxiety and depression.

SECONDARY OUTCOMES:
prevalence and impact of frailty | baseline
  Frailty will be assessed using the Rockwood Clinical Frailty Scale. With scores ranging from 1-9, with higher scores indicating higher frailty.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to third publication — https://pubmed.ncbi.nlm.nih.gov/36870223/
- See also: Link to second publication — https://pubmed.ncbi.nlm.nih.gov/36342627/
- See also: Link to HRA summary of results — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/impact-of-covid-19-on-lung-cancer-patients/